CLINICAL TRIAL: NCT02978365
Title: Factors Associated With Full Recovery After Surgical Repair of Shoulder Instability - Cross Sectional Study
Brief Title: Factors Associated With Full Recovery After Surgical Repair of Shoulder Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uri Gottlieb (Other)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Uri Gottlieb, Head of Physical Therapy Clinic, Medical Corps, Israel Defense Force
Organization: Medical Corps, Israel Defense Force (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IDF-1702-2016; 0177-16-WOMC (Other: Wolfson Medical Center)
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Chronic Instability of Joint
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients (Experimental): Male patients who undergone shoulder surgery to repair chronic instability (at least 1 shoulder dislocation prior to surgery). Time since surgery will be between 26 and 28 weeks. Patients will go through filling questionnaires and isokinetic strength measurements.
  Interventions: Other: Questionnaires; Device: Isokinetic Strength Measurement

INTERVENTIONS:
Other: Questionnaires — Patients will fill self-reported functional shoulder scales (1. Western Ontario Shoulder Instability index - WOSI, and 2. Disabilities of Arm, Shoulder and Hand questionnaire - DASH), as well as a Fear Avoidance Belief Questionnaire (FABQ).
Device: Isokinetic Strength Measurement — Isokinetic strength will be measured using a Biodex Isokinetic System 4.0 (Shirley, NY)

SUMMARY:
Case control study to evaluate different factors (e.g muscle strength, psychological factors) that are associated with full recovery and functional status 6 months after surgical repair of shoulder instability.

DETAILED DESCRIPTION:
In this study the investigators will try to find correlations between different factors and functional abilities of patients 6 months post shoulder surgery.

Patients will be examined in a single encounter for muscle strength, fear avoidance beliefs and functional abilities.

Functional abilities will be examined using two validated questionnaires:

1. The Western Ontario Shoulder Instability index (WOSI)
2. Disabilities of the Arm, Shoulder and Hand (DASH)

Fear avoidance will be evaluated using the Fear Avoidance Belief Questionnaire (FABQ)

Muscle strength of the rotator cuff muscles will be measured using Biodex Isokinetic system, model 4.

ELIGIBILITY:
Inclusion Criteria:

* 26-28 weeks s/p surgical repair of shoulder instability
* At least 1 shoulder dislocation prior to surgery

Exclusion Criteria:

* Previous surgery in either shoulders
* Any injury in the non-operated shoulder in the last 6 months
* Any history of shoulder dislocation or subluxation in the non-operated shoulder
* Any tendon repair during the surgery.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability index (WOSI) | 26-28 weeks post surgery
  Functional scale

SECONDARY OUTCOMES:
Fear avoidance belief questionnaire (FABQ) | 26-28 weeks post surgery
  Fear avoidance questionnaire
Isokinetic strength | 26-28 weeks post surgery
  Ratios between Internal and External rotation strength in both shoulders
Disabilities of Arm, Shoulder and Hand Questionnaire (DASH) | 26-28 weeks post surgery
  Functional scale

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Gam, M.D, Principal Investigator — Medical Corp, Israel Defense Forces
Locations (1):
- IDF Medical Corp, Zrifin, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be published after statistical analysis only.

REFERENCES:
- [Derived] Gottlieb U, Springer S. Translation and validation of a Hebrew version of the Western Ontario Shoulder Instability index. J Orthop Surg Res. 2019 Aug 1;14(1):245. doi: 10.1186/s13018-019-1289-4. PMID 31370869